CLINICAL TRIAL: NCT05541068
Title: The Role of Bioimpedance Analysis in Overweight and Obese Patients With Acute Heart Failure: A Pilot Study
Brief Title: Bioimpedance in Overweight and Obese Patients With Acute Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PIC172-19_FJD
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided by bioimpedance analysis (Active Comparator): These patients were discharged when dry-weight was achieved according to BIA measurements if there was none clinical condition which justified the hospitalization.
  Interventions: Device: Bioimpedance analysis
- Control arm (Active Comparator): In those patients, BIA parameters were not known by the physician responsible. These patients were discharged when they achieved the euvolemic state based in the criteria of their physician
  Interventions: Device: Bioimpedance analysis

INTERVENTIONS:
Device: Bioimpedance analysis — Bioimpedance analysis to achieve assessments of fluid status, especially dry-weight, was performed with the portable Biomasc touch i8 (MaltronInternationl, Essex, UK).

SUMMARY:
Patients with heart failure (HF) have poor prognosis with high mortality and readmission rates. Diuretic therapy is the usual way of managing congestion, but sometimes is difficult to determine when we have reached euvolemia. Even in overweight and obese patients in which physical examination and usual diagnostic techniques have strong limitations. The aim of this study is to investigate the usefulness of bioelectrical impedance analysis (BIA) in management and treatment of HF in overweight and obese patients.

The study included overweight and obese patients who were admitted with acute decompensated HF. The study population was randomized into two arms: BIA-guided therapy or standard care. Serum electrolytes, kidney functions and natriuretic peptides were followed up during their hospital stay and at 90 days after discharge.

The primary endpoint was development of acute kidney injury (AKI) stage III (AKIN-III) during hospitalization and the main secondary endpoint was the reduction of NT-proBNP (N-terminal pro-B-type natriuretic peptide) levels during hospitalization and within 90 days after discharge.

DETAILED DESCRIPTION:
Design: This study was designed as a single-center, single-blind, randomized controlled trial conducted at Hospital Fundación Jimenez Diaz (Madrid, Spain) from February 2020 to December 2021. It is a pilot study which has the objective of obtaining significant results in order to conduct a major research in the future with the purpose of including broadly the use of BIA in HF management. This study was approved by an institutional review committee and performed under Helsinki Declaration Guidelines. All patients provided written informed consent to participate.

Study Procedures All patients included in the study were measured weight and height at admission, and blood tests with hemogram and serum biochemistry including cardiac biomarkers such as NT-proBNP and troponin I were also ordered.

In the first 24 hours after admission an echocardiogram, a lung ultrasound (LUS) and a BIA were done in all patients. BIA was always performed by nephrologists from our hospital not involved in the patient's clinical care. BIA analysis to achieve assessments of fluid status, especially dry-weight, was performed with the portable Biomasc touch i8 (MaltronInternationl, Essex, UK). During the hospitalization period, blood parameters were measured according to standard clinical practice in all patients, with the condition of taking a blood chemistry including NT-proBNP on the day of discharge.

All patients were followed up for 90 days with a new complete blood test including NT-proBNP.

Eligible patients were randomized into two groups:

* Group I (study arm): included 24 patients who received a diuretic treatment guided by BIA. These patients were discharged when dry-weight was achieved according to BIA measurements if there was none clinical condition which justified the hospitalization.
* Group II (control arm): included 24 patients who received the standard clinical practice. In those patients, BIA parameters were not known by the physician responsible. These patients were discharged when they achieved the euvolemic state based in the criteria of their physician.

Outcomes Given the pilot nature of the study the investigators looked for a feasible, clinically meaningful, in-hospital outcome. Development of acute kidney injury (AKI) during hospitalization, defined as an increase in serum creatinine by >0.5 mg/dL (AKIN classification stage III), was the primary outcome. Patients were followed for at least 3 months after discharge. The first secondary outcome was the percentage of patients who achieved levels of NT-proBNP levels <1.000 pg/mL within 90 days after discharge.

Additional secondary outcomes included length of stay in hospital, NT-proBNP reduction >30% during hospitalization, and the combined endpoint of all-cause death, rehospitalization for HF or visit to the ED (emergency department) because of congestion symptoms measured at 90 days after discharge. Patients were contacted by telephone or returned for hospital or outpatient visits.

Statistical analysis Discrete variables were summarized as counts and percentages. Continuous variables were described using median and interquartile range (IQR)and were tested for normality using the Kolmogorov-Smirnov or Shapiro-Wilk test.Baseline characteristics were compared among standard treatment vs BIA-guided treatment with the chi-square test or Fisher´s test for discrete variables, and with Student´s t test and non-parametric Mann-Whitney test for normally and non-normally distributed quantitative variables respectively. Primary and secondary outcomes were also compared between both treatment groups using a chi-square test for independence.Results of these analyses were considered exploratory to study future differences between the groups in terms of time to first adverse outcome or event-free survival. A two-sided P value of less than 0.05 was considered to be statistically significant for all analyses. All statistical analyses were performed using SPSS for Windows Version 19.0 (IBM Corp, Armonk NY).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for Acute Heart Failure (first episode or decompensation), based on Framingham criteria and NT-ProBNP>300 pg/ml
* Body mass index greater than or equal to 25 kg/m2 at admission.

Exclusion Criteria:

* Hemodynamic instability,
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) <15 ml/min/1.73m2, Pregnancy,
* Amputated patients,
* Chronic treatment with corticosteroids,
* Severe valvular heart disease with indication for intervention,
* Dementia or life-expectancy of 1 year or less with high probability for noncompliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Development of acute kidney injury | Through hospitalization, an average of 7 days
  Rate of patients with acute kidney injury (AKI) during hospitalization, defined as an increase in serum creatinine by >0.5 mg/dL (AKIN classification stage III)

SECONDARY OUTCOMES:
levels of NT-proBNP levels <1.000 pg/mL | 90 days after discharge.
  Percentage of patients who achieved levels of NT-proBNP levels <1.000 pg/mL within 90 days after discharge.
Length of stay in hospital. | Through hospitalization, an average of 7 days
  Length of stay in hospital.
NT-proBNP reduction >30% during hospitalization | Through hospitalization, an average of 7 days
  Rate of patients with NT-proBNP reduction >30% during hospitalization
The combined endpoint of all-cause death, rehospitalization for HF or visit to the ED because of congestion symptoms measured at 90 days after discharge | 90 days after discharge.
  The combined endpoint of all-cause death, rehospitalization for HF or visit to the ED

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maria Pello, MD, PhD, Principal Investigator — Fundacion Jimenez Diaz University Hospital, IIS-FJD
Locations (1):
- Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz, Madrid, Spain